CLINICAL TRIAL: NCT06154200
Title: A Pilot Randomized Controlled Trial of Eyelid Androgen Treatment in Dry Eye
Brief Title: Eyelid Androgen Treatment in Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Southern California College of Optometry at Marshall B. Ketchum University (Other)
Responsible Party: Principal Investigator, Jerry Paugh, Professor, Southern California College of Optometry at Marshall B. Ketchum University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-18
Record Dates: First submitted 2023-11-20; First posted 2023-12-04 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Aqueous Tear Deficiency; Meibomian Gland Dysfunction of Bilateral Eyes (Disorder)
Keywords: testosterone; fluorescein breakup time; androgen; dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Intervention Model Description: Subjects randomized to either placebo or drug
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vehicle Gel (Placebo Comparator): Vehicle gel applied to eyelids twice per day
  Interventions: Drug: Vehicle gel
- Testosterone gel 4.5% (Active Comparator): Testosterone gel 4.5% applied to eyelids twice per day
  Interventions: Drug: Testosterone gel 4.5%

INTERVENTIONS:
Drug: Testosterone gel 4.5% — Testosterone gel applied to eyelids twice per day
  Other Names: androgen gel 4.5%
  Arms: Testosterone gel 4.5%
Drug: Vehicle gel — Vehicle gel applied to eyelids twice per day
  Other Names: placebo
  Arms: Vehicle Gel

SUMMARY:
The purpose of this research study is to evaluate the effectiveness and safety of applying androgen sex hormone (i.e., testosterone) gel on the eyelids in the treatment of dry eye patients. Several studies have demonstrated positive treatment effects in dry eye, but few have applied testosterone gels to the eyelids.

DETAILED DESCRIPTION:
The purpose of this study is to examine the safety and efficacy of transdermal eyelid application of testosterone gel along with the length of any beneficial effect following cessation of treatment.

Moderate to severe dry eye subjects will be enrolled into a randomized controlled trial with assignment to either an ~ 4.5% FDA-approved androgen gel (Natesto®, Acerus Pharmaceuticals, Mississagua, Canada) or a placebo formulated similar to Natesto® without testosterone. The gel will be applied to both eyelids in the morning and 12 hours later on both eyelids for a 30 day treatment period

Subjects will fulfil DEWS II criteria for eligibility and further be classified as moderate or severe based on DEWS II recommendations. A standardized examination involving signs and symptoms of dry eye and monitoring function of the meibomian and lacrimal glands, as well as clinical tear and ocular surface measures, IOP, and serum testosterone levels, at baseline, following 30 days of testosterone application, and at one and two months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe dry eye (TBUT < 6.0 seconds, corneal staining > grade 1.5, evidence of meibomian gland secretion compromise or Schirmer < 5 mm wetting in 5 minutes)
* Age over 18
* Mild ectropion
* Previous contact lens wearers IF no wear for prior 6 months
* Punctal plugs if more than three months since placement
* Systemic tetracyclines, antihistamines if consistent dosing
* Sjogren's syndrome and related autoimmune conditions can be enrolled
* Patients using topical dry eye treatments (e.g., Restasis) if willing to discontinue for 30 days

Exclusion Criteria:

* If artificial tears or autologous serum used on day of study
* Ocular surgery if less than 12 months
* Punctal plugs if within 3 months of plug insertion
* Contact Lens wear within the six months prior to study
* PSA levels greater than 4 ng/ml or BPH
* Recent or current thrombolism
* Recent or current cardiovascular events (e.g., MI, stroke)
* Recent or current liver disorders
* Concurrent use of topical medications; e,g., topical glaucoma medications
* Diabetics
* Females of child-bearing age if not on reliable birth control
* History of breast cancer
* Cannot be taking insulin, warfarin or systemic corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-04-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Paugh, OD, PhD, Principal Investigator — SCCO at MBKU
Locations (1):
- Southern California College of Optometry at Marshall B. Ketchum University, Fullerton, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle Gel | Testosterone Gel 4.5%
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Gel | Testosterone Gel 4.5% | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (14.6) | 52.9 (11.3) | 52.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 9 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Fluorescein tear breakup time [Mean (Standard Deviation); unit: seconds] — time in seconds for tear breakup to occur
  seconds | 3.3 (0.9) | 3.6 (1.2) | 3.5 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Tear Break up Time
Description: Time to first dark spot appearance in the tear film
Time Frame: From baseline to 4 weeks treatment
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: eyes
Arm/Group | Vehicle Gel | Testosterone Gel 4.5%
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 12 | 12
seconds | 0.0 (1.2) | 2.9 (1.3)

2. Secondary Outcome: Lower Meibomian Gland Secretion Score (0 - 32 Scale)
Description: 8 central lower meibomian glands are evaluated using gentle (vs forceful) expression. Each secretion is given a score of 0 (clear normal meibum), 1 (cloudy low viscosity) 2 (thick, opaque, 3 inspissated or 4 (no secretion visible). One-half scale increments are used.
Time Frame: From baseline to 4 weeks treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Vehicle Gel | Testosterone Gel 4.5%
Number analyzed (Participants) | 12 | 12
Number analyzed (eyes) | 12 | 12
units on a scale | 0.7 (0.3) | 5.5 (2.1)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Vehicle Gel | Testosterone Gel 4.5%
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT06154200/Prot_SAP_002.pdf
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT06154200/ICF_004.pdf